CLINICAL TRIAL: NCT05672121
Title: A Phase I/II, Open-label, Multiple-cohort, Dose-escalation Study to Evaluate the Safety and Tolerability of KH631 Gene Therapy in Subjects With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Safety and Tolerability of KH631 Gene Therapy in Subjects With Neovascular Age-related Macular Degeneration (nAMD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Origen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KH631-40101
Record Dates: First submitted 2022-12-21; First posted 2023-01-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- KH631 Dose 1 (Experimental): dose1:Administered by Subretinal injection. Dosage form: injection solution. Dose: 200uL. Frequency of administration: one time injection.
  Interventions: Drug: KH631
- KH631 Dose 2 (Experimental): dose2:Administered by Subretinal injection. Dosage form: injection solution. Dose: 200uL. Frequency of administration: one time injection.
  Interventions: Drug: KH631
- KH631 Dose 3 (Experimental): dose3:Administered by Subretinal injection. Dosage form: injection solution. Dose: 200uL. Frequency of administration: one time injection.
  Interventions: Drug: KH631
- KH631 Dose 4 (Experimental): dose4:Administered by Subretinal injection. Dosage form: injection solution. Dose: 200uL. Frequency of administration: one time injection.
  Interventions: Drug: KH631
- KH631 Dose 5 (Experimental): dose5:Administered by Subretinal injection. Dosage form: injection solution. Dose: 200uL. Frequency of administration: one time injection.
  Interventions: Drug: KH631

INTERVENTIONS:
Drug: KH631 — KH631: AAV vector containing a coding sequence for an anti-VEGF protein

SUMMARY:
KH631 is a adeno-associated virus (AAV) vector-based gene therapy for subretinal injection. The long-term, stable therapeutic protein after one time injection for nAMD could potentially reduce the treatment burden and maintain vision.

ELIGIBILITY:
Inclusion Criteria:

* 1.Are willing and able to sign the study written informed consent form (ICF); 2. Men and women ≥ 50 and ≤85 years of age, diagnosed with nAMD at the Screening visit; 3. Subjects must be under active anti-VEGF treatment for nAMD and received a minimum of 3 injections within 6 months prior to screening; 4. Response to anti-VEGF therapy(Response is defined as reduction in CRT≥50μm or at least 30% reduction in fluid by OCT compared to disease at the worst); 5. BCVA between ≤20/63 and ≥20/400(≤63 and ≥19 Early Treatment Diabetic Retinopathy Study [ETDRS] letters) for the first patient in each cohort followed by BCVA between ≤20/40 and ≥20/400(≤73 and ≥19 ETDRS letters) for the rest of the cohort; 6. Must be pseudophakic(at least 3 months after intraocular lens implantation) in the study eye; 7.Female subjects must have been postmenopausal for at least 1 year.

Exclusion Criteria:

* 1.Any other cause of CNV, including pathologic myopia, etc, or other diseases except nAMD have an influence on the test of macular or affect the central visual acuity; 2.Presence of an implant, refractive media opacity affects fundus examination or narrow pupil of the study eye; 3.Active or history of retinal detachment in the study eye; 4.Uncontrolled glaucoma or ocular hypertension; 5.Have taken the drug known to have retinal toxicity; 6.History of intraocular surgery; 7.Uncontrolled hypertension despite medication at the screening visit.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Safety | 24 weeks
  incidence of AEs and SAEs
Change in best corrected visual acuity | 52 weeks
  BCVA

SECONDARY OUTCOMES:
Safety | 104 weeks
  incidence of AEs and SAEs
Change in best corrected visual acuity | 104 weeks
  BCVA
Change in central retinal thickness | 104 weeks
  CRT
Change in area of retinal leakage | 104 weeks
  Leakage measured by FFA
Rescue injections | 104 weeks
  Mean number of rescue injections

OTHER OUTCOMES:
KH631 protein in aqueous fluid and blood | 104 weeks
  Exploratory
VEGF-A in aqueous fluid and blood | 104 weeks
  Exploratory

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wei, PhD, Principal Investigator — Beijing Tongren Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No